CLINICAL TRIAL: NCT02657005
Title: A Phase 1 / 2, Dose Escalation Study of Intravenous TK216 in Patients With Relapsed or Refractory Ewing Sarcoma
Brief Title: TK216 in Patients With Relapsed or Refractory Ewing Sarcoma
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Sponsor Decision
Sponsor: Oncternal Therapeutics, Inc (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TK216-01
Record Dates: First submitted 2016-01-12; First posted 2016-01-15 (Estimated); Results first posted 2024-11-07 (Actual); Last update posted 2025-02-12 (Actual); Status verified 2025-01

CONDITIONS: Sarcoma, Ewing
MeSH Terms: conditions — Sarcoma, Ewing

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- TK216 treatment (Experimental): Dose escalation and expansion cohorts to determine dose-limiting toxicities, maximally tolerated dose, preliminary efficacy, and recommended phase 2 dose.
  Interventions: Drug: TK216

INTERVENTIONS:
Drug: TK216 — Inhibitor of protein-protein interactions of EWS-FLI1 fusion protein

SUMMARY:
Ewing sarcoma is characterized by genomic rearrangements resulting in over-expression of ets family transcription factors driving tumor progression. TK216 is designed to inhibit this effect by inhibiting downstream effects of the EWS-FLI1 transcription factor. This study is a first in human study of TK216 in subjects with Ewing sarcoma. The study is designed to establish initial safety and efficacy data in monotherapy and in combination with vincristine to assess the potential of TK216 for further development.

DETAILED DESCRIPTION:
The study has been expanded to explore single agent TK216 for longer treatment duration. Approximately 26 patients will be enrolled in this Cohort.

Please note: This study has been terminated and is no longer enrolling patients.

ELIGIBILITY:
1. Major Inclusion Criteria (for all Study Parts or protocol versions unless specifically noted):

Patients who meet the following inclusion criteria will be eligible to participate in this study:

1. Willing and able to provide written IRB/IEC-approved Informed Consent. For patients < 18 years of age, their parent or legal guardian must sign a written informed consent. Assent, when appropriate, will be obtained according to institutional guidelines.
2. Have histologically or cytologically confirmed diagnosis of Ewing sarcoma (including ESFT) with relapsed or refractory disease

   1. who have failed standard therapy and for whom no known curative therapy exists (For Parts 1-3), OR
   2. patients with metastatic disease who had standard chemotherapy at the time of diagnosis (For Part 4) (NOTE: as of Protocol version 7, pathology reports and slides or blocks should be available for review or additional testing. If not available, site must discuss with Sponsor.)
3. Measurable disease according to RECIST version 1.1. Measurable disease can be verified from a previously documented CT scan or MRI as long as no anti-cancer treatments have been administered in the interim.
4. Must have a central venous catheter in place prior to initiating infusion of study drug.
5. Prior cancer therapy:

   1. Patients may have received any number of prior therapy regimens (For Parts 1-3) OR
   2. Patients may have received no more than 5 prior systemic regimens. At the time of treatment initiation, at least 2 weeks or 5 half-lives, whichever is longer, must have elapsed since prior cytotoxic chemotherapy. At least 7 days must have elapsed since completion of any prior non-cytotoxic cancer therapy (For Part 4).
6. Prior radiotherapy is allowed

   1. If ≥ 2 weeks have elapsed for local palliative XRT (small port); ≥ 6 months must have elapsed if prior total body irradiation, craniospinal XRT or if > 50% radiation of the pelvis; > 6 weeks must have elapsed if other substantial bone marrow radiation. Patients who have received brain irradiation must have completed whole brain radiotherapy and/or gamma knife at least 4 weeks prior to enrollment (For Parts 1-3) OR
   2. If ≥ 4 weeks has elapsed for radiation therapy (RT); ≥ 6 months must have elapsed if prior total body irradiation, craniospinal RT or if > 50% radiation of the pelvis; > 6 weeks must have elapsed if other substantial bone marrow radiation. Patients who have received brain irradiation must have completed whole brain radiotherapy and/or gamma knife at least 4 weeks prior to enrollment (For Part 4).
7. Stem Cell Transplant or Rescue without TBI: No evidence of active graft vs. host disease and ≥ 3 months must have elapsed since transplant.
8. Patients with controlled asymptomatic CNS involvement are allowed.
9. Eastern Cooperative Oncology Group (ECOG) performance status (PS) ≤ 2 in patients ≥17 years old; or Karnofsky/Lansky >50 in patients <16 years old.
10. Age:

    a. Cohort 1: Patient's age >18 years old. b. Cohorts 2-6: Patients must be > 12 years old. c. Cohorts 7-10: Patients must be ≥ 10 years old. d. Cohort 11: Patient's age ≥ 8 years (For Part 4)
11. Life expectancy of at least 3 months.
12. Adequate organ function as measured by baseline laboratory values. 13. Cardiac ejection fraction > 50% or shortening fraction > 28%. 14. Females of child-bearing potential must have a negative pregnancy test (within 7-days of starting treatment) during screening and subjects must be willing to use effective contraception. be neither breastfeeding nor intending to become pregnant during study participation. Females of childbearing potential must agree to avoid pregnancy during the study and commit to abstinence from heterosexual intercourse or agree to use two methods of birth control (one highly effective method and one additional effective method) at least 4 weeks before the start of protocol therapy, for the duration of study participation, and for 6 months after the last dose of TK216. 15. Males with partner(s) of childbearing potential must take appropriate precautions to avoid fathering a child from the screening period until 90 days after receiving the last dose of TK216. They must commit to abstinence from heterosexual intercourse or agree to use appropriate barrier contraception.

16. Willingness and ability to comply with scheduled visits, treatment plan, laboratory tests and other study procedures.

Major Exclusion Criteria:

Patients will not be enrolled if they meet any one of the following exclusion criteria:

1. Current participation in another therapeutic clinical trial.
2. Symptomatic brain metastases.
3. History of previous cancer (non ES), except squamous cell or basal-cell carcinoma of the skin or any in situ carcinoma that has been completely resected, which required therapy within the previous 3 years.
4. Any of the following in the past 6 months: symptomatic congestive heart failure, cerebrovascular accident or transient ischemic attack, pulmonary embolism, deep vein thrombosis, symptomatic bradycardia, requirement for antiarrhythmic medication.
5. History of prolonged QTc interval (e.g., repeated demonstration of a QTc interval > 450 milliseconds, unless associated with the use of medications known to prolong the QTc interval). (NOTE: For Part 4, repeated demonstration of a QTc interval > 470 milliseconds) 6. History of additional risk factors for torsade de pointes (e.g., heart failure, family history of long QT syndrome

7. Use of concomitant medications that increase or possibly increase the risk to prolong the QTc interval and/or induce torsades de pointes ventricular arrhythmia.

8. Females who are breastfeeding/lactating. 9. Known active infections (bacterial, fungal, viral including hepatitis and HIV positivity). 10. Other severe acute or chronic medical or psychiatric condition or laboratory abnormality that may increase the risk associated with study participation or study drug administration or may interfere with the interpretation of study results and, in the judgment of the Investigator, would make the patient inappropriate for entry into this study or could compromise protocol objectives in the opinion of the Investigator and/or the Sponsor.

Min Age: 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 85 (Actual)
Dates: Start 2016-08 (Actual); Primary Completion 2022-05 (Actual); Study Completion 2022-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: James Breitmeyer, MD, Study Director — Oncternal Therapeutics
Locations (9):
- United States (9):
  - UCLA Jonsson Comprehensive Cancer Center, Los Angeles, California
  - Children's Hospital of Colorado, Aurora, Colorado
  - Children's National Hospital, Washington D.C., District of Columbia
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Duke Cancer Institute, Durham, North Carolina
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Oregon Health & Science University, Portland, Oregon
  - Texas Children's Cancer & Hematology Centers, Baylor College, Houston, Texas
  - UT MD Anderson Cancer Center, Houston, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Meyers PA, Federman N, Daw N, Anderson PM, Davis LE, Kim A, Macy ME, Pietrofeso A, Ratan R, Riedel RF, Trucco M, Breitmeyer JB, Toretsky JA, Ludwig JA. Open-Label, Multicenter, Phase I/II, First-in-Human Trial of TK216: A First-Generation EWS::FLI1 Fusion Protein Antagonist in Ewing Sarcoma. J Clin Oncol. 2024 Nov;42(31):3725-3734. doi: 10.1200/JCO.24.00020. Epub 2024 Jul 2. PMID 38954782

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 85 subjects were enrolled in this study across eight North American centers. The pathologic diagnoses were confirmed at each enrolling center. Most patients were heavily pretreated, with the median number of prior therapies being 3.0 (range, 1-10). The gender and ethnicity of the enrolled patients matched ES's prevalence in the U.S. population.
Pre-assignment Details: Once an appropriate patient has been identified, a 30-day screening period began and evaluated eligibility.
  The study was executed in several Parts:
  Part 1: Dose Escalation Segment (Cohorts 1-6) Part 2: Schedule Escalation Segment (Cohorts 7-9) Part 3: Expansion Segment (Cohort 10) Part 4: Dose and Schedule Evaluation Segment (Cohort 11)
  Note: For purposes of result summaries, Cohorts 1-8 pooled, Cohorts 9 & 10 pooled, and Cohort 11 will be displayed.
Groups:
- 18 mg/m^2 (7 Days); 36 mg/m^2 (7 Days); 72 mg/m^2 (7 Days); 144 mg/m^2 (7 Days); 200 mg/m^2 (10 Days); 200 mg/m^2 (14 Days): Dose Escalation Segment (Cohorts 1-6) was an open label, "3+3" patient enrollment scheme, sequential allocation, dose finding allocation of the sequential allocation of TK216 monotherapy. The length of TK216 infusion for all dose escalation cohorts was 7 days. A lower intermediate dose of 220mg/m2 /day for 7 days was determined to be the maximum tolerated dose (MTD) for the 7-day continuous infusion of TK216.
- 220 mg/m^2 (7 Days); 220 mg/m^2 (10 Days); 288 mg/m^2 (7 Days): Schedule Escalation Segment (Cohorts 7-9) was an open label, "3+3" patient enrollment scheme, sequential allocation of the increase in length of infusion of TK216 monotherapy. Following the first two cycles, vincristine could be added as tolerated up to 2mg on the first day of each cycle. The recommended Phase 2 dose (RP2D) was determined to be 200mg/m2 /day for 14 days followed by a 14-day recovery period, per 28-day cycle
- Expansion Cohort: Expansion Segment (Cohort 10) where patients were treated with the schedule for RP2D of TK216 with vincristine 0.75 - 1.5 mg/m2 administered on the first day of each 28-day cycle
- 175 mg/m^2 (28 Days): Dose and Schedule Evaluation Segment (Cohort 11) where patients received a starting dose of 175mg/m2 /day of TK216 intravenously by continuous infusion for 28 days per cycle. If the patient's tumor response was determined by the Investigator as inadequate after at least one protocol-specified post-baseline assessment and they were not experiencing toxicities at this dose level, the Investigator could increase the dose to 200 mg/m2/day after discussion with the Sponsor. Vincristine (0.75 to 1.5 mg/m2 up to a maximum dose of 2 mg) could be administered in parallel with the TK216 infusion following progressive disease after TK216-01 monotherapy but only after consultation with the Sponsor.
Period: Overall Study
Arm/Group | 18 mg/m^2 (7 Days) | 36 mg/m^2 (7 Days) | 72 mg/m^2 (7 Days) | 144 mg/m^2 (7 Days) | 200 mg/m^2 (10 Days) | 200 mg/m^2 (14 Days) | 220 mg/m^2 (7 Days) | 220 mg/m^2 (10 Days) | 288 mg/m^2 (7 Days) | Expansion Cohort | 175 mg/m^2 (28 Days)
Started | 3 | 3 | 3 | 3 | 4 | 4 | 3 | 3 | 7 | 44 | 8
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 3 | 3 | 3 | 3 | 4 | 4 | 3 | 3 | 7 | 44 | 8

BASELINE CHARACTERISTICS:
Population: Safety Population
Groups:
- Total: Total of all reporting groups
Arm/Group | 18 mg/m^2 (7 Days) | 36 mg/m^2 (7 Days) | 72 mg/m^2 (7 Days) | 144 mg/m^2 (7 Days) | 200 mg/m^2 (10 Days) | 200 mg/m^2 (14 Days) | 220 mg/m^2 (7 Days) | 220 mg/m^2 (10 Days) | 288 mg/m^2 (7 Days) | Expansion Cohort | 175 mg/m^2 (28 Days) | Total
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 4 | 4 | 3 | 3 | 7 | 44 | 8 | 85
Age, Continuous [Mean (Standard Deviation); unit: years] | 28.0 (5.3) | 38.7 (28.7) | 41.3 (12.7) | 33.3 (10.7) | 30.0 (9.5) | 25.5 (7.9) | 24.7 (8.1) | 24.0 (10.0) | 23.7 (6.3) | 29.2 (14.6) | 27.0 (10.0) | 28.9 (13.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 3 | 1 | 0 | 0 | 1 | 2 | 1 | 2 | 16 | 2 | 29
  Male | 2 | 0 | 2 | 3 | 4 | 3 | 1 | 2 | 5 | 28 | 6 | 56
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 5 | 1 | 0 | 7
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 2
  Black or African American | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  White | 3 | 2 | 3 | 2 | 4 | 4 | 3 | 2 | 0 | 41 | 5 | 69
  More than one race | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 4
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 2 | 3

OUTCOME MEASURES:

1. Primary Outcome: Overall Response Rate
Description: Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1) for target lesions and assessed by MRI: Complete Response (CR), Disappearance of all target lesions and pathologic lymph nodes; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions, no new lesions, and no progression of non-target lesions; Overall Response (OR) = CR + PR.
Time Frame: 36 months
Population: All Patients
Measure: Count of Participants; unit: Participants
Arm/Group | 18 mg/m^2 (7 Days) | 36 mg/m^2 (7 Days) | 72 mg/m^2 (7 Days) | 144 mg/m^2 (7 Days) | 200 mg/m^2 (10 Days) | 200 mg/m^2 (14 Days) | 220 mg/m^2 (7 Days) | 220 mg/m^2 (10 Days) | 288 mg/m^2 (7 Days) | Expansion Cohort | 175 mg/m^2 (28 Days)
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 4 | 4 | 3 | 3 | 7 | 44 | 8
Participants | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0

ADVERSE EVENTS:
Time Frame: Treatment emergent adverse events were collected from first treatment received through end of study for all patients. (i.e., 36 months)
Description: Per clinicaltrials.gov definitions
Groups:
- Expansion: Expansion Segment (Cohort 10) where patients were treated with the schedule for RP2D of TK216 with vincristine 0.75 - 1.5 mg/m2 administered on the first day of each 28-day cycle
- 175 mg/m^2: Dose and Schedule Evaluation Segment (Cohort 11) where patients received a starting dose of 175mg/m2 /day of TK216 intravenously by continuous infusion for 28 days per cycle. If the patient's tumor response was determined by the Investigator as inadequate after at least one protocol-specified post-baseline assessment and they were not experiencing toxicities at this dose level, the Investigator could increase the dose to 200 mg/m2/day after discussion with the Sponsor. Vincristine (0.75 to 1.5 mg/m2 up to a maximum dose of 2 mg) could be administered in parallel with the TK216 infusion following progressive disease after TK216-01 monotherapy but only after consultation with the Sponsor
Arm/Group | 18 mg/m^2 (7 Days) | 36 mg/m^2 (7 Days) | 72 mg/m^2 (7 Days) | 144 mg/m^2 (7 Days) | 200 mg/m^2 (10 Days) | 200 mg/m^2 (14 Days) | 220 mg/m^2 (7 Days) | 220 mg/m^2 (10 Days) | 288 mg/m^2 (7 Days) | Expansion | 175 mg/m^2
All-Cause Mortality (participants affected / at risk) | 2/3 | 2/3 | 3/3 | 3/3 | 4/4 | 2/4 | 2/3 | 3/3 | 3/7 | 26/44 | 1/8
Serious Adverse Events (participants affected / at risk) | 1/3 | 1/3 | 1/3 | 1/3 | 4/4 | 1/4 | 2/3 | 1/3 | 2/7 | 21/44 | 5/8
Other Adverse Events (participants affected / at risk) | 3/3 | 3/3 | 3/3 | 3/3 | 4/4 | 4/4 | 3/3 | 3/3 | 7/7 | 44/44 | 8/8
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 18 mg/m^2 (7 Days) (N=3) | 36 mg/m^2 (7 Days) (N=3) | 72 mg/m^2 (7 Days) (N=3) | 144 mg/m^2 (7 Days) (N=3) | 200 mg/m^2 (10 Days) (N=4) | 200 mg/m^2 (14 Days) (N=4) | 220 mg/m^2 (7 Days) (N=3) | 220 mg/m^2 (10 Days) (N=3) | 288 mg/m^2 (7 Days) (N=7) | Expansion (N=44) | 175 mg/m^2 (N=8)
Febrile Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (3) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 4 (4) | 2 (2)
Abdominal Pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Hypercalcaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Aortobronchial fistula (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Device Related Infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Hypoglossal nerve paralysis (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haematemesis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cancer Pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Skin Infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Periorbital cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Influenza like illness (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (3) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pericardial effusion (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (5) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cardiopulmonary failure (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
COVID-19 (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Bacteremia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (4) | 0 (0)
Device dislocation (Product Issues) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Jugular vein thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Blood Creatinine increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pain in jaw (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pleuritic Pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Catheter site cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Complication associated with device (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | 18 mg/m^2 (7 Days) (N=3) | 36 mg/m^2 (7 Days) (N=3) | 72 mg/m^2 (7 Days) (N=3) | 144 mg/m^2 (7 Days) (N=3) | 200 mg/m^2 (10 Days) (N=4) | 200 mg/m^2 (14 Days) (N=4) | 220 mg/m^2 (7 Days) (N=3) | 220 mg/m^2 (10 Days) (N=3) | 288 mg/m^2 (7 Days) (N=7) | Expansion (N=44) | 175 mg/m^2 (N=8)
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 3 | 2 | 0 | 3 | 4 | 26 | 6
Anaemia (Blood and lymphatic system disorders) | 0 | 1 | 2 | 2 | 4 | 1 | 0 | 3 | 4 | 22 | 5
Leukopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 2 | 2 | 0 | 3 | 4 | 18 | 2
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 2 | 2 | 0 | 0 | 2 | 3 | 6 | 4
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 2 | 3 | 4 | 2
Fatigue (General disorders) | 0 | 0 | 1 | 2 | 2 | 2 | 1 | 3 | 3 | 18 | 1
Pyrexia (General disorders) | 0 | 2 | 1 | 1 | 2 | 2 | 1 | 3 | 3 | 15 | 1
Nausea (Gastrointestinal disorders) | 1 | 1 | 0 | 0 | 1 | 1 | 0 | 2 | 2 | 16 | 1
Constipation (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 2 | 2 | 0 | 2 | 9 | 2
Diarrhoea (Gastrointestinal disorders) | 1 | 0 | 0 | 1 | 1 | 1 | 1 | 0 | 3 | 6 | 1
Abdominal Pain (Gastrointestinal disorders) | 1 | 1 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 5 | 1
Lymphocyte cunt decrease (Investigations) | 1 | 0 | 0 | 0 | 3 | 2 | 0 | 0 | 1 | 5 | 2
Blood creatinine increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 4 | 0
Weight decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 5 | 0
Back Pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 8 | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 6 | 3
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 1 | 5 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 5 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 1 | 3 | 6 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 0 | 2 | 0 | 0 | 1 | 0 | 0 | 0 | 4 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 3 | 0
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 5 | 0
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 3
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 3 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 3 | 0 | 2 | 2 | 16 | 3
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 3 | 2 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1 | 0 | 3 | 0 | 1 | 0 | 9 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 1 | 4 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 3 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 3 | 0
Headache (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 2 | 1 | 2 | 1 | 13 | 1
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 4 | 0
Paraesthesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 5 | 0
Bacteraemia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 1
Sinus tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 1 | 5 | 0
Tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 4 | 0

LIMITATIONS AND CAVEATS:
TK216 was advanced as a novel inhibitor of EWS::FLI1 despite pharmacologic challenges to creating an oral formulation. In vivo studies showed that continuous exposure to TK216 was required for optimal efficacy.47 This continuous infusion was a logistical challenge and negatively affected study enrollment rates. Another limitation of this study was the lack of a pharmacodynamic readout of TK216 activity.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-07-20): https://cdn.clinicaltrials.gov/large-docs/05/NCT02657005/Prot_SAP_000.pdf